CLINICAL TRIAL: NCT04633239
Title: A Phase 1/1b Dose Escalation Study of Abemaciclib and Olaparib for Recurrent Platinum-Resistant Ovarian Cancer
Brief Title: Testing the Addition of Abemaciclib to Olaparib for Women With Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-10084; NCI-2020-10084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10422 (Other: Yale University Cancer Center LAO); 10422 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma
MeSH Terms: interventions — abemaciclib; Biopsy; Specimen Handling; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abemaciclib, olaparib, biospecimen collection) (Experimental): Patients receive olaparib PO BID on days 1-28 and abemaciclib PO BID on days 8-28 of cycle 1 and days 1-28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and undergo tumor biopsy on study.
  Interventions: Drug: Abemaciclib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Olaparib

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY 2835219; LY-2835219; LY2835219; Verzenio
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase I/Ib trial identifies the side effects and best dose of abemaciclib when given together with olaparib in treating patients with ovarian cancer that responds at first to treatment with drugs that contain the metal platinum but then comes back within a certain period (recurrent platinum-resistant). Abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Olaparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep tumor cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. Adding abemaciclib to olaparib may work better to treat recurrent platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of abemaciclib plus olaparib in patients with platinum-resistant ovarian cancer by determining the maximum tolerated dose and recommended phase 2 dose.

SECONDARY OBJECTIVE:

I. To observe and record anti-tumor activity using overall response rate (ORR) and duration of response (DoR) with abemaciclib and olaparib, given in combination, in patients with platinum-resistant ovarian cancer.

EXPLORATORY OBJECTIVES:

I. To assess proof of mechanism (RB, phosphoRB, cleaved caspase 3, Ki67, geminin, gamma-H2AX, RAD51 nuclear foci, pNBS multiplex, Myc transcriptional targets ODC1 and LDHA, homologous recombination genes BRCA1, BRCA2, RAD51, serum thymidine kinase), plasma and tumor pharmacokinetics, and subgroups of response (immunohistochemistry [IHC] for Myc, cyclin E; next generation sequencing [NGS]/whole exome sequencing [WES] for DCAF, hormone receptor [HR] repair gene alterations, Myc, and CCNE1; ribonucleic acid sequencing [RNAseq] for Myc and CCNE1).

II. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

III. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Experimental Therapeutics Clinical Trials Network (EET) Biobank at Nationwide Children's Hospital.

OUTLINE: This is a dose-escalation study of abemaciclib.

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28 and abemaciclib PO BID on days 8-28 of cycle 1 and days 1-28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and undergo tumor biopsy on study.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed recurrent platinum-resistant epithelial ovarian carcinoma (EOC) of any histology, as defined by progression within 6 months of the last dose of platinum-based chemotherapy. Both primary platinum resistant and acquired platinum resistant patients are allowed
* High-grade serous histology is required (for the dose expansion cohort only) (data on BRCA (e.g. germline BRCA, Somatic BRCA, Neither, Unknown) and homologous recombination deficiency (HRD)/Loss of Heterozygosity (LOH) (e.g. HRD > 42/LOH >16%, HRD score < 42/LOH < 16%, Unknown) is not required for study but will be collected if available
* Patients must have received 1-3 prior systemic therapies
* Women age >= 18 years. Because no dosing or adverse event data are currently available on the use of abemaciclib in combination with olaparib in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 10 g/dL (within 28 days prior to administration of study treatment)

  * Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion
* Absolute neutrophil count >= 1,500/mcL (within 28 days prior to administration of study treatment)
* Platelets >= 100,000/mcL (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)

  * Patients with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN, unless liver metastases are present in which case they must be =< 5 x ULN (within 28 days prior to administration of study treatment)
* Patients must have creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation or based on a 24-hour urine test (within 28 days prior to administration of study treatment)
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2 (within 28 days prior to administration of study treatment). Estimated GFR calculated using Cockcroft-Gault equation
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Patients with treated brain metastases are eligible if patient is stable for at least 4 weeks status post (s/p) radiation therapy and off corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the screening period
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Postmenopausal or evidence of non-childbearing status, a negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50
  * Radiation-induced oophorectomy with last menses > 1 year ago
  * Chemotherapy-induced menopause with > 1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* The effects of abemaciclib and olaparib on the developing human fetus are unknown. For this reason and because CDK-and PARP-inhibiting agents are known to be teratogenic, women of child-bearing potential and their partners, who are sexually active, must agree to the use of one highly effective form of contraception and their partner must use a male condom prior to study entry, for the duration of study participation, and for 6 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* For the dose expansion cohort, patients must have disease amenable to biopsy for correlative studies, specifically at least 1 tumor accessible and safe for biopsy on office exam or tumor that a radiologist deems is safe for biopsy in interventional radiology department based on imaging (dose expansion cohort only). For the dose escalation cohort, patients with evaluable disease are acceptable
* For inclusion in i) the optional genetic research and ii) the optional biomarker research, patients must fulfill the following criteria:

  * Provision of informed consent for genetic research prior to collection of sample
  * Provision of informed consent for biomarker research prior to collection of sample
  * If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study
* Patients may not have received prior CDK 4/6 inhibitors. Previous PARP inhibitor use is allowed in front-line treatment but not for recurrent disease
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] grade =< 1) from the acute effects of chemotherapy except for residual alopecia or grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy)
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 28 days is required between end of radiotherapy and randomization
* For agents other than chemotherapy, a 4 week washout period is required. Previous bevacizumab use is allowed
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* History of allergic reaction or hypersensitivity attributed to compounds of similar chemical or biologic composition to abemaciclib, olaparib or any of the excipients of these products
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because abemaciclib is a CDK-inhibiting agent and olaparib is a PARP inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with abemaciclib and olaparib, breastfeeding should be discontinued if the mother is treated with abemaciclib and olaparib
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT [QTcF] prolongation > 500 ms, electrolyte disturbances, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest, etc.), or patients with congenital long QT syndrome
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML)
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection that, in the judgment of the investigator, would preclude participation in this study. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance < 30 ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea)
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients with an active systemic fungal infection
* Patients with suspected or history of interstitial lung disease (ILD)/pneumonitis
* Patients with active thromboembolism. Active thromboembolism is defined as a diagnosis of a thromboembolic within the last 6 months or continued evidence of thromboembolism on imaging despite stable anti-coagulation for 6 months. Patients with a history of thromboembolism > 6 months ago on anti-coagulation as continued prevention are eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | 28 days (end of cycle 1)
  Safety and tolerability will be measured using Common Terminology Criteria for Adverse Events (CTCAE) version 5. The number of patients experiencing a dose limiting toxicity will be tabulated. The recommended phase 2 dose will be determined by the dose escalation phase using 3+3 design.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 30 days after completion of study treatment
  ORR will be calculated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of response (DoR) | 30 days after completion of study treatment
  DoR will be calculated using RECIST version 1.1. The duration of overall response is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

OTHER OUTCOMES:
Biomarker analysis | 30 days after completion of study treatment
  Will measure proof of mechanism (RB, phosphoRB, cleaved caspase 3, Ki67, geminin, gamma-H2AX, RAD51 nuclear foci, pNBS multiplex, Myc transcriptional targets ODC1 and LDHA, homologous recombination genes BRCA1, BRCA2, RAD51, serum thymidine kinase), plasma and tumor pharmacokinetics, and subgroups of response (immunohistochemistry [IHC] for Myc, cyclin E; next generation sequencing [NGS]/whole exome sequencing [WES] for DCAF, hormone receptor [HR] repair gene alterations, Myc, and CCNE1; ribonucleic acid sequencing [RNAseq] for Myc and CCNE1).

CONTACTS AND LOCATIONS:
Overall Officials: Camille Jackson, Principal Investigator — Yale University Cancer Center LAO
Locations (27):
- United States (27):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm